CLINICAL TRIAL: NCT02583815
Title: Feasibility of Activity Monitoring in Patients With Cancer: Physical Activity Monitoring in Cancer Patients (PAMCap)
Acronym: PAMCap
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: STU 062015-021
Record Dates: First submitted 2015-10-20; First posted 2015-10-22 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Gastrointestinal Cancer; Breast Cancer; Gynecologic Cancer; Genitourinary Cancer; Leukemia; Lung Cancer; Skin Cancer; Endocrine Cancer; Male Genital Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms; Breast Neoplasms; Urogenital Neoplasms; Leukemia; Lung Neoplasms; Skin Neoplasms; Endocrine Gland Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected at each study visit (Baseline, then every weeks until week 12 (+/-14 days). Prior to storage, complete the sample inventory logs for each subject so that specimen chain of custody can be established. Samples will be frozen at -80°C until the time of analysis.
  Include in each shipment batch copies of: 1) the blood collection source documents for each patient; and 2) copies of each subjects specimen inventory form
  Keep originals of these documents in the subject's chart
  Samples will be analyzed using a multiplexed ELISA method (Meso Scale Discovery) for IL-1beta, IL-6, IL-10 and TNF-alpha
  With explicit participant consent, samples will also be processed for DNA and stored for future analysis.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Cancer Patients: This is an open label feasibility pilot study of commercially available physical activity monitoring devices in patients receiving systemic therapy at the Harold Simmons Cancer Center, UT Southwestern Medical Center.

SUMMARY:
This is an open label feasibility pilot study of commercially available physical activity monitoring devices in patients receiving systemic therapy at the Harold Simmons Cancer Center, UT Southwestern Medical Center.

DETAILED DESCRIPTION:
Study will be conducted for 12 weeks (+/-14 days) of monitoring.

BASELINE ASSESSMENTS Baseline assessment should be performed within 14 days of Week 1.

1. Signed informed consent;
2. ECOG Performance Status per treating physician (chart abstraction of available data);
3. Pathology report confirming cancer diagnosis;
4. Psychosocial assessment questionnaires;
5. Blood for correlative biomarkers (10 ml);
6. Documentation of planned/ongoing chemotherapy regimen

ON-STUDY ASSESSMENTS

1. Physical Activity Monitor (PAM)

   1. Fitbit (PAM) devices will be provided by investigators for the period of the study;
   2. Introduction to the device and instructions on use and care will be provided based on commercial marketing material;
   3. Subjects will be assisted in setting up Fitbit device on smart phone;
   4. Subjects will be asked to wear Fitbit device continuously for 12 weeks - however, the device should not be worn during bathing or showering;
   5. Subjects will be asked to sync their Fitbit devices to the database at least once a week;
   6. Clinical coordinator may send phone or text reminders to encourage syncing as Fitbit device can only record 1 weeks' worth of data;
   7. Cost Coverage
   8. Investigators will purchase devices prior to start of study with grant funding.
   9. PAM Accountability
   10. Investigator and investigator site are responsible for maintaining accurate inventory and accountability logs for the devices.
   11. Subjects will be asked to sign a form upon receipt and return of device as applicable.
2. ECOG - Eastern Cooperative Oncology Group Performance Status 0 - Fully active, able to carry on all pre-disease performance without restriction; 1 - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2 - Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours; 3 - Capable of only limited self-care, confined to bed or chair more than 50% of waking hours; 4 - Completely disabled -- cannot carry on any self-care. Totally confined to bed or chair; 5 - Dead
3. Functional Assessment of Cancer Therapy - General (FACT-G).

   a. The FACT-G is a 27-item scale designed to measure multidimensional quality of life in breast cancer patients.
4. Quick Inventory of Depressive Symptomatology - Self-Rated (QIDS-SR116) .

   a. The QIDS-SR16 is a 16-item version of the 30-item Inventory of Depressive Symptomatology (IDS) designed to assess severity of depression-specific symptoms.
5. Pittsburgh Sleep Quality Index (PSQI) (See Appendix H).9

   a. The PSQI is a 19-item scale designed to assess sleep quality and disturbances.
6. Brief Fatigue Inventory (BFI) (See Appendix I).10

   a. The BFI is a 9-item scale designed to assess fatigue in cancer patients.
7. Biomarker and DNA Blood Tests

   1. Blood samples will be collected at each study visit indicated by the study calendar. Process samples according to the sample processing instructions. Prior to storage, complete the sample inventory logs for each subject so that specimen chain of custody can be established. Samples will be frozen at -80°C until the time of analysis;
   2. Include in each shipment batch copies of: 1) the blood collection source documents for each patient; and 2) copies of each subjects specimen inventory form;
   3. Keep originals of these documents in the subject's chart;
   4. Samples will be analyzed using a multiplexed ELISA method (Meso Scale Discovery) for IL-1beta, IL-6, IL-10 and TNF-alpha;
   5. With explicit participant consent, samples will also be processed for DNA and stored for future analysis.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age 18 or above
* Receiving or planning to receive outpatient therapy for any cancer
* Baseline ECOG status 0-2;
* Speak and understand English as all Psychological assessment tools included in this study have not been validated in Spanish;
* Access to smartphone device compatible to sync with PAM Device

Exclusion Criteria:

* Recent injury which may result in impaired mobility;
* Major surgery within 4 weeks or till recovery to baseline functioning (per patient) whichever is shorter;
* Inability to comply with study requirement;
* Medical, psychiatric condition which in the investigators opinion will affect the successful completion of study;
* Current use of a wearable PAM device as defined by use of PAM device in the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving systemic therapy at the Harold Simmons Cancer Center, UT Southwestern Medical Center.
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2015-08; Primary Completion 2017-09-15 (Actual); Study Completion 2017-09-15 (Actual)

PRIMARY OUTCOMES:
Number of Participants Who Use PAM Device | Week 6 until week 12
  The primary endpoint of the study is the feasibility defined by subjects who use a PAM device for more than 42 of 84 days in the observation period (12 weeks +/- 14 days)

SECONDARY OUTCOMES:
Number of Steps | 12 Weeks (+/- 14 days)
  The number of steps will be collected over the course of 12 weeks to help determine the amount of physical activity is being done. The Physical activity monitor is able to track this.
Distance Walked | 12 Weeks (+/- 14 days)
  The distance walked will be collected over the course of 12 weeks to help determine the amount of physical activity is being done. The Physical activity monitor is able to track this.
Time Spent in Activity | 12 Weeks (+/- 14 days)
  The time spent in Activity will be collected over the course of 12 weeks to help determine the amount of physical activity is being done. The Physical activity monitor is able to track this.
Eastern Cooperative Oncology Group Performance Status | Baseline and every 4 weeks for 12 weeks (+/-14 days)
  ECOG assessment data will be extracted by the research team from the Electronic Medical Record.
Functional Assessment of Cancer Therapy. (FACT-G) | Baseline and every 4 weeks for 12 weeks (+/-14 days)
  The FACT-G is a 27-item (self-assessment)scale designed to measure multidimensional quality of life in breast cancer patients.
Quick Inventory of Depressive Symptomatology (QIDS-SR) | Baseline and every 4 weeks for 12 weeks (+/-14 days)
  The QIDS-SR16 is a 16-item (self assessment) version of the 30-item Inventory of Depressive Symptomatology (IDS) designed to assess severity of depression-specific symptoms.
Pittsburgh Sleep Quality Index (PSQI) | Baseline and every 4 weeks for 12 weeks (+/-14 days)
  The PSQI is a 19-item (self assessment) scale designed to assess sleep quality and disturbances.
Brief Fatigue Inventory (BFI) | Baseline and every 4 weeks for 12 weeks (+/-14 days)
  The BFI is a 9-item (self assessment) scale designed to assess fatigue in cancer patients.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Beg, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States